CLINICAL TRIAL: NCT04414683
Title: Factors Affecting the Prognosis of Early Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 109058-E
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: staging surgery — laparoscopic or laparotomic staging surgery

SUMMARY:
To elucidate factors affecting survival of early stage ovarian cancer

DETAILED DESCRIPTION:
To analyze factors affecting survival of early ovarian cancer, such as cell type, cell grade, intraoperative rupture, and laparoscopy vs. laparotomy, etc.

ELIGIBILITY:
Inclusion Criteria:

* early stage ovarian cancer

Exclusion Criteria:

* Nil.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ovarian cancer
Study Population: patients with early stage ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Factors affecting overall survival of early ovarian cancer | 10 years

SECONDARY OUTCOMES:
Factors affecting progression-free survival of early ovarian cancer | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan